CLINICAL TRIAL: NCT01540994
Title: Phase I/II Trial of Stereotactic Hypofractionated Radiotherapy of the Prostate
Brief Title: Stereotactic Body Radiation Therapy (SBRT) for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Responsible Party: Principal Investigator, Geoffrey Weinstein, M.D., Medical Director, Radiation Oncology, Sharp HealthCare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101091
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Prostatic Neoplasm
Keywords: Neoplasms; Urogenital neoplasm; Genital neoplasms, male
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Urogenital Neoplasms; Genital Neoplasms, Male | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Radiotherapy: phase 1/2 (but no drug, biological/vaccine or combination product used)
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Body Radiation Therapy (Experimental): Stereotactic Body Radiation Therapy
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Stereotactic Body Radiation Therapy

SUMMARY:
The purpose of this study is to evaluate a short course (five radiation treatments) of very focused ("stereotactic") external beam radiation therapy for the treatment of early stage prostate cancer.

DETAILED DESCRIPTION:
External beam radiation therapy for prostate cancer, while effective, takes up to 9 weeks to deliver on a Monday through Friday basis. Recent phase I/II studies from Seattle and Palo Alto using stereotactic guidance to deliver high doses of radiation to the prostate over a 1 to 2 week period of time suggest that outcomes may be equal or superior to standard approaches. These data, combined with markedly improved convenience for patients, make radiosurgery (SBRT) for early-stage prostate cancer an enticing option. The goal of this study is to offer a radiosurgical option to patients within the Sharp system under the umbrella of an IRB-approved study.

ELIGIBILITY:
Inclusion Criteria:

* Male with any age (typically 50 to 70 years old) with a low risk disease. This is defined as a Gleason's score of 6 or less, clinical stage of T2a or less, and a PSA of less than 15. We will also include patients with Gleason's score of 3+4=7 if there are fewer than 2 cores positive, with no more than 5mm of tumor in aggregate dimension.

Exclusion Criteria:

* Prior surgery or radiotherapy for prostate cancer, PSA over 10, Gleason scores 7, 8, 9, or 10 (except Gleason 7 as noted, above), or clinical stage T2b, T2c, T3, or T4.

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Weinstein, M.D., Principal Investigator — Sharp HealthCare
Locations (1):
- Sharp Memorial Hospital, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 2011 and 2018 patients with prostate cancer were enrolled from the Radiation Oncology clinic.
Groups:
- Radiation Therapy: Stereotactic Body Radiation Therapy: All patients entered in the study will be referred to the Radiation Oncology department for standard consultation for a newly-diagnosed prostate cancer. During the course of the initial consultation the patients will be given various treatment options depending on their tumor characteristics. If appropriate they will also be given the option of being treated on-protocol using the stereotactic body radiosurgery approach. All patients enrolled on this protocol will receive 35Gy in 5 fractions delivered every other day using a multi-field 6MV photon IMRT technique treating the prostate with limited (2-4mm) margin, and daily rectal balloon placement to assist with prostate immobilization.
Period: Overall Study
Arm/Group | Radiation Therapy: Stereotactic Body Radiation Therapy
Started | 12 (2011)
Completed | 12 (2018)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Between 2011 and 2018, 12 patients were enrolled and received treatment as per protocol specifications.
Groups:
- Radiation Therapy: Prostate Stereotactic Body Radiation Therapy: All patients entered in the study will be referred to the Radiation Oncology department for standard consultation for a newly-diagnosed prostate cancer. During the course of the initial consultation the patients will be given various treatment options depending on their tumor characteristics. If appropriate they will also be given the option of being treated on-protocol using the stereotactic body radiosurgery approach. All patients enrolled on this protocol will receive 35Gy in 5 fractions delivered every other day using a multi-field 6MV photon IMRT technique treating the prostate with limited (2-4mm) margin, and daily rectal balloon placement to assist with prostate immobilization.
Arm/Group | Radiation Therapy: Prostate Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants] — Population: 12 patients received treatment as per protocol specifications.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 5
    >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Acute and Late Genitourinary and Lower Gastrointestinal Toxicity Using the Radiation Therapy Oncology Group Acute and Late Morbidity Scales.
Description: Acute and late genitourinary and lower gastrointestinal toxicity will be evaluated using the Radiation Therapy Oncology Group Acute and Late Morbidity Scales, which range from 0-5, where a high score corresponds to a worse outcome/worse toxicity. Toxicity will be measured weekly during radiation, and every 6-12 months following radiation through patient interview. The acute toxicity score will be defined as the highest score obtained from measurements taken during radiation for each participant. The late toxicity score will be defined as the highest score obtained from measurements taken following completion of radiation for each participant.
Time Frame: Assessed weekly during radiation (from day 1 up to 3 weeks) for acute toxicity, and every 6-12 months following completion of radiation (from 3 weeks up to 84 months) for late toxicity.
Population: 12 participants who were enrolled in the study
Measure: Number; unit: participants
Arm/Group | Radiation Therapy: Prostate Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 12
participants
  Acute Genitourinary Toxicity: 0 (none) | 11
  Acute Genitourinary Toxicity Grade 1 | 0
  Acute Genitourinary Toxicity Grade 2 | 0
  Acute Genitourinary Toxicity Grade 3 | 0
  Acute Genitourinary Toxicity Grade 4 | 1
  Acute Genitourinary Toxicity Grade 5 | 0
  Acute Lower Gastrointestinal Toxicity: 0 (none) | 12
  Acute Lower Gastrointestinal Toxicity Grade 1 | 0
  Acute Lower Gastrointestinal Toxicity Grade 2 | 0
  Acute Lower Gastrointestinal Toxicity Grade 3 | 0
  Acute Lower Gastrointestinal Toxicity Grade 4 | 0
  Acute Lower Gastrointestinal Toxicity Grade 5 | 0
  Late Genitourinary Toxicity: 0 (none) | 8
  Late Genitourinary Toxicity Grade 1 | 4
  Late Genitourinary Toxicity Grade 2 | 0
  Late Genitourinary Toxicity Grade 3 | 0
  Late Genitourinary Toxicity Grade 4 | 0
  Late Genitourinary Toxicity Grade 5 | 0
  Late Gastrointestinal Toxicity: 0 (none) | 10
  Late Gastrointestinal Toxicity Grade 1 | 0
  Late Gastrointestinal Toxicity Grade 2 | 2
  Late Gastrointestinal Toxicity Grade 3 | 0
  Late Gastrointestinal Toxicity Grade 4 | 0
  Late Gastrointestinal Toxicity Grade 5 | 0

2. Secondary Outcome: Rate of Biochemical Disease-free Status
Description: Patients will be followed after completion of treatment with PSA tests every 6-12 months Patients will be deemed to have "biochemical failure" if the post-treatment PSA increases by 2 ng/ml or more above the post-radiation nadir PSA. Patients who do not qualify as having "biochemical failure" will be deemed as "biochemically disease-free".
Time Frame: mean 41 months (range 3-84 months)
Population: 12 participants who were enrolled in the study
Measure: Number; unit: participants
Arm/Group | Radiation Therapy: Prostate Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 12
participants | 10

ADVERSE EVENTS:
Time Frame: Assessed weekly during radiation (from day 1 up to 3 weeks) for acute toxicity, and every 6-12 months following completion of radiation (from 3 weeks up to 84 months) for late toxicity.
Arm/Group | Radiation Therapy: Prostate Stereotactic Body Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy: Prostate Stereotactic Body Radiation Therapy (N=12)
Rectal bleeding (Gastrointestinal disorders) | 1 (1) — One patient hospitalized for rectal bleeding after completion of XRT, but colonoscopy showed diverticulitis without evidence of radiation changes.
Acute Genitourinary Toxicity (Grade 4) (Renal and urinary disorders) | 1 (1) — Bladder outlet obstruction requiring temporary foley catheter placement.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy: Prostate Stereotactic Body Radiation Therapy (N=12)
Late Genitourinary Toxicity (Grade 1) (Renal and urinary disorders) | 4 (4) — Frequency of urination or nocturia twice pretreatment habit/dysuria, urgency not requiring medication
Late Gastrointestinal Toxicity (Grade 2) (Gastrointestinal disorders) | 2 (2) — Moderate diarrhea and colic; bowel movement > 5 times daily; excessive rectal mucus or intermittent bleeding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT01540994/Prot_000.pdf